CLINICAL TRIAL: NCT05249504
Title: Efectividad de la intervención AMICOPE Para Mejorar y/o Mantener la Salud Autopercibida y la Capacidad intrínseca en Personas Mayores: un Ensayo clínico Aleatorizado (EFICIS)
Brief Title: Effectiveness of AMICOPE Intervention to Maintain Self-Perceived Health and Intrinsic Capacity in Older People
Acronym: EFICIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FSIEPI2100537; PI21/00537 (Other Grant/Funding Number: FIS); 5876 (Other: CEEAH UAB)
Record Dates: First submitted 2021-12-15; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Mobility; Depressive Symptoms; Nutrition, Healthy; Cognitive Decline; Hearing Loss; Visual Impairment
Keywords: Frailty; Intrinsic capacity; Multicomponent intervention; Randomized clinical Trial; Quality of life
MeSH Terms: conditions — Depression; Cognitive Dysfunction; Hearing Loss; Vision Disorders; Frailty | interventions — Nutritional Status; Psychology; Personal Autonomy; Community Resources

STUDY DESIGN:
Intervention Model Description: Open and Pragmatic Parallel Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Intervention group (Experimental): AMICOPE multicomponent intervention:
  * Physical activity (VIVIFRAIL program): 10 hours.
  * Nutrition: 6,5 hours.
  * Psychology: 6,5 hours.
  * Personal autonomy: 4,5 hours
  * Learn about community resources: 2, 5 hours
  Interventions: Other: VIVIFRAIL; Other: Nutrition; Behavioral: Psychology; Behavioral: Personal autonomy; Other: Community resources
- 2. Control group (Active Comparator): Control group participants will receive usual advice on healthy lifestyle habits and a follow-up phone call from healthcare professionals.
  Interventions: Other: Standard recommendations

INTERVENTIONS:
Other: VIVIFRAIL — VIVIFRAIL is a set of physical activity programs (designed according to several elderly functional level profiles) aimed to prevent motor disability and improve quality of life. It works endurance, flexibility, balance and strength.
  https://web.archive.org/web/20210907041944/https://vivifrail.com/
  Arms: 1. Intervention group
Other: Nutrition — Sessions to learn about personal nutrition habits, offer nutritional advice, and acquire skills to incorporate simple healthy nutrition guidelines into everyday life. A visit to a supermarket to make it easier to read and understand the basic information on nutrition labels.
  Arms: 1. Intervention group
Behavioral: Psychology — Relaxation techniques to manage mood, a photo-elicitation dynamic to address loneliness, and a dynamic to collectively develop a map of health assets in the neighborhood or territory to obtain information on community resources. Finally, a group visit is planned to a community facility previously agreed upon by the participants.
  Arms: 1. Intervention group
Behavioral: Personal autonomy — Review practical cases on personal autonomy, the proper use of medications, and discover basic cognitive stimulation strategies.
  Arms: 1. Intervention group
Other: Community resources — Learn about community resources
  Arms: 1. Intervention group
Other: Standard recommendations — Usual advice provided at primary care office accompanied to booklets about healthy lifestyles
  Arms: 2. Control group

SUMMARY:
In their day to day, persons do from simple to more or less complicated tasks and activities (ie: stand from a chair, open a door, shopping, read, drive, play chess, remind an appointment...). Such ability to do things is called capacity. Intrinsic capacity is the combination of all the physical and mental capacities that a person has, and reach its maximum in the early adulthood and then declines as the person ages. Each kind of capacity declines at her own speed (which may be faster or slower according to each person lifestyle), and once drops below a threshold may lead to a reduction in quality of life and loss of autonomy.

Nevertheless there are some actions that may be effective to prevent or slow such decline. To do so the investigators have design an intervention that combines several things of different nature (what is know as a complex intervention) called AMICOPE. The AMICOPE intervention is performed in the community or in primary care centers through 12 weekly group sessions of 2 h 30 min which combine structured and adapted physical activity, group dynamics to promote social support and address loneliness, social isolation and depressive symptoms, and dietary advice.

Our study is addressed to persons over 70 with light problems in mobility, nutrition or mood state.

The purpose of this study is to assess if the AMICOPE intervention is better than the standard advice to follow healthy lifestyles to improve or maintain self-perceived health, mobility, nutritional status an psychological wellbeing.

ELIGIBILITY:
INCLUSION CRITERIA

* To live in the community
* To be able to move autonomously to the intervention place
* To Have a deficit in at least one mobility, vitality or psychological domains in the Integrated Care for Older People (ICOPE) screening tool confirmed by a reference test, namely:

A - Mobility: unable to stand up from a chair 5 times in less than 14 seconds AND having less than 10 points in the Short Physical Performance Battery (SPPB).

B - Vitality: any nutritional problem from the ICOPE screening tool (loss of appetite OR losing more than 3 Kg not intentionally in the last 3 months) AND having less than 12 points in MNA (malnutrition or malnutrition risc).

C - Psychological: any depressive symptoms from the ICOPE screening tool (answer that in the last two weeks has had feelings of sadness, melancholy OR hopelessness or refer lack of interest or pleasure when doing things) AND the presence of at least two or more symptoms on the 5-item Geriatric Depression Scale (GDS5).

EXCLUSION CRITERIA

* People with previous diagnosis of dementia or cognitive decline with a score below 24 points in the Minimental State Examination (MMSE).
* People in the end of life.
* People who have factors that prevent or contraindicate the performance of the planned interventions, such as contraindication to physical activity, mental or (non-corrected) communication issues that makes it difficult to participate in group dynamics.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-perceived health | Baseline, after the intervention (average 16 weeks)
  Change in self-perceived health status according to the Euroqol Visual Analogue Scale, where participants scores from 0 (worse state) to 100 (better state) their current perceived health

SECONDARY OUTCOMES:
Functional status | Baseline, after the intervention (average 16 weeks)
  Change in functional status according to the Short Physical Performance Battery (SPPB), a set of tests that measure balance, gait speed and strength (raising 5 times from a chair). Persons are classified in categories according to their final score (0-3, 4-6, 7-9, 10-12). Higher scores indicates robustness, lower scores are indicative of frailty and disability.
Nutritional status | Baseline, after the intervention (average 16 weeks)
  Change in nutritional risks assessed by the abridged version of Mini-Nutritional Assessment (MNA), which classifies the persons as normal (12-14 points), at risk of malnutrition (8-11) or malnourished (0-7)
Depressive symptoms | Baseline, after the intervention (average 16 weeks)
  Change in proportion of participants with depressive symptoms using the 5 items Geriatric Depression Scales (GDS5). Not depressed (0 or 1 point), Depressed (2-5).
Autonomy in daily life. | Baseline, after the intervention (average 16 weeks)
  Change in the ability to perform basic and instrumental daily life activities will be measured with the Short-Form Late-Life Function and Disability Instrument (SF-LLFDI).
  Higher scores indicates a higher level of autonomy.
Health related quality of life. | Baseline, after the intervention (average 16 weeks)
  Change in health related quality of life will be assessed with the quality of life questionnaire EQ-5D-5L.
Physical activity. | Baseline, after the intervention (average 16 weeks)
  Change in level of physical activity, which will be assessed with the Spanish Short Version of the Minnesota Leisure Time Physical Activity Questionnaire (VREM), which according to the time doing several activities computes the energy expenditure in units that can be compared between them, the Metabolic Equivalent of Task. (MET). Persons are categorized as sedentary (< 1.250 METs-min/14 days), moderately active (1.250 to 2.999 METs-min/14 days); active (3.000 to 4.999 METs-min/14 days) or very active (≥ 5.000 METs-min/14 days).)
Loneliness | Baseline, after the intervention (average 16 weeks)
  Change in the degree of Loneliness, which will be assessed with De Jong Gierveld Loneliness Scale. The degree of loneliness is scored as no loneliness (0 to 2 points), mild loneliness ( 3 to 8), severe (9 to 10) or very severe (11)
Social support and risk of isolation | Baseline, after the intervention (average 16 weeks)
  Change in social support and risk of isolation, which will be assessed with the Lubben Social Network Scale - Revised (LSNS-R). According the the LSNS-R score the persons will be classified as with low risk (30 to 60 points); mild (26 to 30); high (21 to 25) or socially isolated (0 to 20).

IPD SHARING:
Plan to Share IPD: Yes
The sponsor only will share data from participants that have provided written consent to share its anonymized data for studies with scientific purposes related with well-being, quality of life and autonomy of the elderly persons.
  Once the database is closed all identifying data collected to develop the study (ie: names and contact phones to make appointments) will be removed from the database.
  Any date variable will be replaced by a time reference variable, taking as reference the day of the first visit (ie: instead of date of birth and date of visit, will be replaced by the age).
  Other actions may be performed to ensure a reasonable balance between the data loss and the risk of re-identification, as editing quasi-identificatory variables (ie categorizing/aggregating participant data, as creating age groups) or removed (ie removing the data identifying the centers) or removing cases with a high degree of singularity given the quasi-identificatory variables combination.
Time Frame: The data can be requested 18 months after publishing the results.
Access Criteria: Upon request by non-profit organizations. The purpose of the request must match the purpose for which the participants have given their sharing consent.
  Requester must cite and recognize the source of the data in their works, as far as the funds that the project has received.